CLINICAL TRIAL: NCT02586103
Title: Prospective Study Assessing the Validity of Y-PAS (Yale Preoperative Anxiety Scale) to Predict Patients Undergoing Magnetic Resonance Imaging Without the Use of Sedation/General Anesthesia
Status: Completed | Type: Observational
Sponsor: Arlyne Thung (Other)
Responsible Party: Sponsor-Investigator, Arlyne Thung, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00894
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI: Patients who undergo simulated practice MRI on the day of or prior to their scheduled MRI.
  Interventions: Device: MRI simulation

INTERVENTIONS:
Device: MRI simulation — It is not a working MRI machine but sounds and feels just like the real machine.

SUMMARY:
The mYPAS (Modified Yale Preoperative Anxiety Scale) is a quick, easy, validated and "gold standard" assessment tool to measure pediatric anxiety in the perioperative period. Therefore the objective of the current prospective study is examine if the mY-PAS is an effective screening tool to differentiate patients who would succeed versus fail for MRI without sedation/anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* all patients and parents who are willing to participate in the simulated practice MRI on the day of or prior to their scheduled MRI.

Exclusion Criteria:

* patients/parents who refuse to go through the practice MRI sessions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for MRI with sedation or anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Anxiety score | Immediately following MRI simulation
  Modified Yale Preoperative Anxiety Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States